CLINICAL TRIAL: NCT06097078
Title: Prospective, Multi-centre, Exploratory and Observational One-arm Study to Evaluate Preemptive Endoluminal Vacuum Therapy to Prevent Anastomotic Leakage After Esophagectomy Due to Esophageal Cancer
Brief Title: Endoluminal Vacuum Therapy to Prevent Anastomotic Leakage After Esophagectomy Due to Esophageal Cancer
Acronym: ESPY
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2209
Record Dates: First submitted 2023-10-16; First posted 2023-10-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Cancer; Esophagus Cancer; Anastomotic Leak
Keywords: endoluminal vacuum therapy; anastomotic leakage; esophagectomy; esophageal cancer; abdominal and cardiac surgery
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eso-SPONGE®: endoluminal vacuum therapy to prevent anastomotic leakage after esophagectomy due to esophageal cancer
  Interventions: Device: Eso-SPONGE®

INTERVENTIONS:
Device: Eso-SPONGE® — minimally invasive treatment and prevention of anastomotic leakages and perforations in the upper gastrointestinal tract (upper GIT)
  Other Names: endoluminal vacuum therapy (EVT) device

SUMMARY:
A prospective, multi-centre, exploratory and observational one-arm study to evaluate preventive Endoluminal Vacuum Therapy(pEVT) to prevent anastomotic leakage after esophagectomy due to esophageal cancer. The main objective is to evaluate the potential protective effect of prophylactic preemptive endoluminal vacuum therapy on esophageal-gastric anastomosis dehiscence after esophagectomy.

DETAILED DESCRIPTION:
Prospective, multi-centre, exploratory and observational one-arm study to evaluate preemptive endoluminal vacuum therapy to prevent anastomotic leakage after esophagectomy due to esophageal cancer.

The study comprises a maximum of 5 visits per protocol. At visit 0, informed consent will be obtained, and the patient will be checked for compliance with all inclusion criteria and no exclusion criteria in the study. Demographic characteristics, medical history and oncological parameters will be collected. At visit 1 ttMILE will be carry out and immediately (0-24h) after completion of the anastomosis, in patients who meet selection criteria, the Eso-SPONGE® will be placed endoscopically via an overtube, as usual clinical practice of the centre. The tube will be routed transnasally and then connected to a vacuum pump, generating a continuous negative pressure of 75 mmHg. The Eso-SPONGE system will be checked 6-hourly for leakage and dislocation. The sponge will be removed after 4-6 days (V2). After removal, the anastomosis and the gastric tube will be assessed endoscopically to exclude leakage and evaluate ischemia and stenosis, and the pylorus will be evaluated for spasm. The next visits (V3 and V4) will be carried out at 30 and 90 days after the intervention has been placed. Leakage, ischemia and stenosis will be clinically evaluated at each visit and a new endoscopy will be performed in patient who show symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for total minimally invasive (laparoscopic or robotic and thoracoscopic) transthoracic Ivor Lewis esophagectomy (ttMILE) due to esophageal cancer and subsequent eso-SPONGE application to prevent anastomotic leakage
* Patients able to read and understand the Patient Information Sheet and sign, if accepted, the Informed Consent Form
* Patients able, at the discretion of the investigator, to comply with the requirements of the study and without impediments to follow the instructions and assessments throughout the study.

Exclusion Criteria:

* Patients undergoing transhiatal esophagectomy without reconstruction, open Ivor Lewis esophagectomy or other esophageal resections different to ttMILE.
* Multi-organ resection during the esophagectomy.
* Emergent-urgent esophagectomy.
* Coloplasty or small bowel plasty.
* Necrotic tissue/gangrene.
* Blood clotting disorder.
* Bleeding esophageal varices.
* Sponge placement required directly on major vessels.
* Patients with known sensitivities or allergies to its components
* Participation in any other clinical trial and use of any drug or experimental device, currently or in the 4 weeks prior to inclusion in the study.
* Women who are pregnant, suspected of being pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a total minimally invasive (laparoscopic or robotic and thoracoscopic) transthoracic Ivor Lewis esophagectomy (ttMILE) due to esophageal cancer and subsequent eso-SPONGE® application to prevent anastomotic leakage (AL)
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with anastomotic leakage | throughout the duration of the study (until last follow-up at postoperative day 90)
  Anastomotic leakage (AL) is a severe complication following gastric and esophageal surgery. Anastomotic leakage occurs in 5-30% of patients after esophagectomy and may be further complicated by mediastinitis, sepsis, multiple organ failure, or death. The primary objective of the study is to evaluate the potential protective effect of prophylactic preemptive endoluminal vacuum therapy on esophageal-gastric anastomosis dehiscence after esophagectomy.

SECONDARY OUTCOMES:
Comprehensive Complication Index | Postoperative day 30 and day 90
  The Comprehensive Complication Index (CCI®) calculates the overall morbidity of a patient after any surgical intervention based on the complication grading by the "Clavien-Dindo Classification" (CDC). The Comprehensive Complication Index (CCI®) reflects the gravity of this overall complication burden on the patient on a scale from 0 (no complication) to 100 (death).
Description of Adverse Events | throughout the duration of the study (until last follow-up at postoperative day 90)
  All the Adverse Events reported during the study will be described together with their characteristics, noting those related with the investigational device application.
Rate of postoperative ischemia | Postoperative day 30 and day 90
  The different grades of postoperative ischemia at Visit 1, Visit 2 and Visit 3
Rate of postoperative mortality | Postoperative day 30 and day 90
  The percentage of patients who died along the study will be described in terms of absolute and relative frequencies, as well as causes for death and time until death regarding investigational device application.
Rate of postoperative stenosis | throughout the duration of the study (until last follow-up at postoperative day 90)
  The percentage of postoperative stenosis at Visit 1, Visit 2 and Visit 3, as well as along the study
Length of hospitalization | until discharge (approximately 10 days postoperatively)
  time elapsed until reaching the "fit for discharge criteria" regarding investigational device application
Re-admissions to hospital | throughout the duration of the study (until last follow-up at postoperative day 90)
  The percentage of patients re-admitted along the study will be described; as well as the time elapsed until re-admission regarding investigational device application
Surgical reoperations | throughout the duration of the study (until last follow-up at postoperative day 90)
  The percentage of patients with surgical reoperations along the study will be described; as well as the time elapsed until surgical reoperation regarding investigational device application
Anastomotic leakage free survival | throughout the duration of the study (until last follow-up at postoperative day 90)
  Event free survival at 30 days and at 90 days will be analyzed using Kaplan-Meier method, considering the anastomotic leakage reported during the study. Patients with no anastomotic leakage during the analyzed period will be censored at last follow-up date
Rate of intraluminal hemorrhage | throughout the duration of the study (until last follow-up at postoperative day 90)
  The percentage of patients with intraluminal hemorrhage along the study will be described in terms of absolute and relative frequencies; as well as the time elapsed until hemorrhage regarding investigational device application. Additionally, to see the distribution of the time until intraluminal hemorrhage Kaplan-Meier method will be performed at 90 days (patients with no intraluminal hemorrhage during the study will be censored at last follow-up date).

CONTACTS AND LOCATIONS:
Overall Officials: Dulce Momblán García, Dr., Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No